CLINICAL TRIAL: NCT01128842
Title: A Phase 1, Open-Label Study Of Neratinib (HKI-272) In Combination With Capecitabine In Japanese Subject With Solid Tumors
Brief Title: A Study Of Neratinib (HKI-272) And Capecitabine In Japanese With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-1122 / B1891018
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Neratinib; Capecitabine; Combination; Solid Tumor
MeSH Terms: interventions — neratinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neratinib + Capecitabine (Experimental): Neratinib + Capecitabine
  Interventions: Drug: Neratinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Neratinib — 240 mg once daily by mouth.
Drug: Capecitabine — 1500 mg/m^2 twice daily by mouth.

SUMMARY:
This is an open-label, phase 1 study of a single cohort of neratinib (HKI-272) in combination with capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 20 years and older
* Confirmed pathologic diagnosis of a solid tumor not curable with currently available therapies, for which neratinib plus capecitabine is a reasonable treatment option.
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Please note: ascites, pleural or pericardial effusion, osteoblastic bone metastases, and carcinomatous lymphangitis of the lung will not be considered measurable lesions).
* Subjects with skin lesions that are measurable by computed tomography (CT) scans or magnetic resonance imaging (MRI) as the only site of measurable disease are allowed.
* Recovery from all clinically significant adverse events (AEs) related to prior therapies (excluding alopecia).
* Left ventricular ejection fraction (LVEF) within institutional range of normal as measured by multi-gated acquisition (MUGA) or echocardiogram (ECHO).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (not declining within 2 weeks before signing the informed consent form [ICF]).

Screening lab values within the following parameters: Absolute neutrophil count (ANC): 1.5×109/L (1500/mm3) Platelet count: 100×109/L (100,000/mm3) Hemoglobin: 9.0 g/dL (90 g/L) Serum creatinine: 01.5×upper limit of normal (ULN) Total bilirubin: 1.5×ULN (<3 ULN if Gilbert's disease) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): 2.5×ULN (=5×ULN if liver metastases are present)

* For women of childbearing potential, a negative urine or serum pregnancy test result before study entry.
* All subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control for the duration of the study and for 28 days after the last dose of investigational product. A subject is biologically capable of having children if he or she is using contraceptives or if his or her sexual partner is sterile or using contraceptives.

Exclusion Criteria:

* Prior treatment with anthracyclines with a cumulative dose of doxorubicin >400 mg/m², or of epirubicin >800 mg/m², or the equivalent dose for other anthracyclines or derivatives.
* Major surgery, chemotherapy, radiotherapy, any investigational agents, or other cancer therapy within at least 2 weeks before administration of the first dose of investigational product.
* Bone as the ONLY site of disease .
* Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (subjects with a history of CNS metastases or cord compression are permitted if they have been definitively treated and are off anticonvulsants and steroids for at least 4 weeks before cycle 1 day 1).

QT (corrected QT (QTc)) interval >0.47seconds or a known history of QTc prolongation or torsades de pointes.

* Presence of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association [NYHA] functional classification of 02), angina requiring treatment, myocardial infarction within the past 12 months, or any clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention.
* Pregnant or breastfeeding women.
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom (eg, Crohn's disease, malabsorption, or grade 2 or higher diarrhea of any etiology at baseline).
* Inability or unwillingness to swallow tablets (neratinib and capecitabine).
* Subjects with active or uncontrolled renal insufficiency, in whom medication dose adjustments are indicated.
* Subject known to be human immunodeficiency virus (HIV) seropositive and/or have acute or chronic hepatitis B infection (hepatitis B surface antigen [HBsAg] positive) or hepatitis C infection (anti-HCV positive).
* Known history of hypersensitivity to capecitabine or any of it components, including 5-FU.
* Any other cancer within 5 years prior to screening with the exception of contralateral breast carcinoma, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin.
* Clinically significant ongoing or recent infection within 2 weeks before administration of the first dose of investigational product.
* Evidence of significant medical illness or abnormal laboratory findings that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study, or preclude the evaluation of the subject's response. Examples include, but are not limited to, serious active infection, (ie, requiring intravenous antibiotic or antiviral agent) or uncontrolled major seizure disorder, significant pulmonary disorder (eg, interstitial pneumonitis, pulmonary hypertension), or psychiatric disorder that would interfere with subject safety or informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (2):
- Japan (2):
  - Investigational Site, Shizuoka
  - Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib + Capecitabine: Neratinib: 240 mg once daily by mouth, Capecitabine: 1500 mg/m^2 twice daily.
Period: Overall Study
Arm/Group | Neratinib + Capecitabine
Started | 7
Completed | 0
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Disease Progression | 6

BASELINE CHARACTERISTICS:
Groups:
- Neratinib + Capecitabine: Neratinib: 240 mg, continuous once daily by mouth Capecitabine: 1500 mg/m^2 twice daily by mouth
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.43 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) - Percentage of Participants With DLT Events
Description: DLT was defined as 1. Grade 3 or 4 non-hematologic toxicity (exceptions listed below as a.-c.), a. Grade 3 asthenia was NOT considered to be a DLT UNLESS it lasted >3 days. b. Grade 3 nausea or vomiting was NOT considered to be a DLT UNLESS the subject was already receiving optimal medical therapy. c. Grade 3 or 4 infection was NOT considered to be a DLT UNLESS it is associated with grade 3 or 4 neutropenia. 2. Grade 3 diarrhea that lasted >2 days while the subject was on optimal medical therapy or that was associated with fever (greater than or equal 38.0 ºC) or grade 3 dehydration. 3. Grade 4 neutropenia lasting ≥3 days or grade 4 febrile neutropenia. 4. Grade 4 thrombocytopenia lasting ≥3 days or complicated with bleeding or requiring platelet transfusion. 5. Delayed recovery (to National Cancer Institute [NCI] grade 1 or less, or baseline) from any of the toxicities listed above (items 1-4), that was related to study drug, and that delayed the next dose by more than 3 weeks.
Time Frame: From first dose date to day 21.
Population: The safety population was defined as all subjects who received at least 1 dose of investigational product (neratinib and/or capecitabine).
Measure: Count of Participants; unit: Participants
Groups:
- Neratinib + Capecitabine: Neratinib: 240 mg once daily by mouth, Capecitabine: 1500 mg/m^2 twice daily by mouth.
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Best Overall Response
Description: Number of participants with Partial Response (PR) or Complete Response (CR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) (v1.0) criteria. CR: Disappearance of all lesions; PR: at least a 30% decrease in the sum of longest diameters (SLD) of target lesions, taking as reference the baseline SLD; Progressive Disease (PD): at least a 20% increase in the SLD of target lesions, taking as reference the nadir longest diameter, meaning the smallest SLDs recorded since the treatment started, or the appearance of 1 or more new lesions, or unequivocal progression of existing nontarget lesions; and stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since treatment started.
Time Frame: From first dose date to progression or last tumor assessment, up to 41 weeks.
Population: All subjects who met Inclusion and Exclusion criteria, received at least 2 weeks of Investigational Product, and underwent at least 1 Follow Up (FU) tumor assessment at approximately cycle 2 (week 6). Subjects who died or had PD including symptomatic deterioration before the scheduled FU tumor assessment were included in the evaluable population.
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
Participants
  Partial Response | 1
  Stable Disease | 4
  Progressive Disease | 2

3. Secondary Outcome: Objective Response Rate
Description: Percentage of participants with partial response (PR) or complete response (CR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: CR, disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; and Non Progressive Disease (PD) for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to 41 weeks.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
percentage of participants | 14.3 [0.40 to 57.9]

4. Secondary Outcome: Progression Free Survival
Description: Number of weeks between the date of the first dose of test article and the first date of disease recurrence or disease progression (PD), or death due to any cause, was documented, censored at the last evaluation, investigator assessment. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (v1.0), as at least a 20% increase in the sum of the longest diameters (LD) of target lesions, taking as reference the nadir LD, meaning the smallest sum of the LDs recorded since the treatment started; or unequivocal progression of existing nontarget lesions; or the appearance of any new lesions.
Time Frame: From first dose date to PD or death, up to 41 weeks.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
weeks | 15.6 [5.4 to 36.1]

5. Secondary Outcome: Area Under the Curve (AUC) of Neratinib in Combination With Capecitabine
Description: AUC of Neratinib at day 14 following Administration of Neratinib 240 mg in combination with Capecitabine 1500 mg/m^2 per day to Japanese Subjects with Cancer.
Time Frame: At 1, 2, 4, 6, 8 and 21-24 hours after dose on day 14.
Population: The pharmacokinetic population was defined as all subjects who received at least 1 dose of investigational product (neratinib and/or capecitabine).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
ng*hr/mL | 1070 (619)

6. Secondary Outcome: Maximum Plasma Concentration of Neratinib in Combination With Capecitabine
Description: Maximum plasma concentration (nanograms/milliliter) of Neratinib at day 14 following Administration of Neratinib 240 mg in combination with Capecitabine 1500 mg/m^2 per day to Japanese Subjects with Cancer.
Time Frame: Measured at 1, 2, 4, 6, 8 and 21-24 hours after dose on day 14.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
ng/mL | 61.9 (32.0)

7. Primary Outcome: Tolerated Dose
Description: Six subjects will be initially enrolled (neratinib 240 mg/day; capecitabine 1500 mg/m²/day on days 1 through 14). AEs and DLTs will be assessed from the first dose of investigational product through day 21. Based on the DLT rate in these first 6 subjects, dose tolerability will be confirmed as follows:
  If ≤1 of the first 6 evaluable subjects experience a DLT by day 21, then this dose is considered tolerable, and enrollment will stop.
  If ≥3 of the first 6 evaluable subjects experience a DLT by day 21, this dose is considered intolerable.
  If 2 of the first 6 evaluable subjects experience a DLT by day 21, then an additional 4 subjects will be enrolled at the same dose level.
  If a total of 10 subjects are enrolled, then the tolerability will be confirmed as follows:
  If ≤3 of the total 10 subjects experience a DLT by day 21, then this dose will be considered tolerable.
  If ≥4 of the total 10 subjects experience a DLT by day 21, then the dose will be considered intolerable.
Time Frame: From first dose date to day 21.
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | Neratinib + Capecitabine
Number analyzed (Participants) | 7
mg | 240

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to 41 weeks.
Arm/Group | Neratinib + Capecitabine
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib + Capecitabine (N=7)
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib + Capecitabine (N=7)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 4
Oesophagitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 5
Mucosal inflammation (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Cystitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 4
Tinea infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less